CLINICAL TRIAL: NCT06665451
Title: Evaluation of Erythropoietin Gel Effect on Stability of Immediate Implant ( Clinical and Radiographical Study )
Brief Title: Erythropoietin Gel Effect on Dental Implant Stability
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Mohsen Farghaly, Principle investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Implant surface modification
Record Dates: First submitted 2024-10-25; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Osseointegration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Group (Experimental): Patients with fresh extraction sockets in the anterior maxilla will be treated by immediate implant coated by erythropoietin gel .
  Interventions: Other: Erythropoietin gel coated implants
- Control group (Active Comparator): Patients with fresh extraction sockets in the anterior maxilla will be treated by non coated immediate implant .
  Interventions: Other: Non coated dental implants

INTERVENTIONS:
Other: Non coated dental implants — Patients with fresh extraction sockets in the anterior maxilla will be treated by non coated immediate implant .
  Arms: Control group
Other: Erythropoietin gel coated implants — Patients with fresh extraction sockets in the anterior maxilla will be treated by immediate implant coated by erythropoietin gel.
  Arms: Test Group

SUMMARY:
* Achieving and maintaining long-term osseointegration for dental implants is a key objective in the field of dentistry. The success of osseointegration is influenced by the surface treatment applied to dental implants. Numerous coating techniques have been developed to improve and speed up osseointegration.
* The aim of the current study is to assess immediate dental implant stability coated with erythropoietin gel, both clinically and radiographically.
* Materials and Methods: We conducted a randomized controlled clinical trial.The sample will include patients demanding immediate implant treatment in the anterior maxilla . Patients will be randomly allocated into the two groups of the study. The group A will be treated with erythropoietin gel coated dental implant immediately after extraction of non restorable teeth in the anterior maxilla . Group B will be treated with non coated dental implant immediately after extraction of non restorable teeth in the anterior maxilla .
* The primary outcome variable will be implant stability and the secondary outcome will be crestal marginal bone level and bone density around implants. It will be measured at time of implant placement and reevaluated after 6-months .

ELIGIBILITY:
Inclusion Criteria:

* All patients Should have nonrestorable teeth in the anterior maxilla indicated for extraction and seeking implant placement.
* Good general periodontal health and maintenance.

Exclusion Criteria:

* Heavy smokers who smoke more than ten cigarettes per day
* Acute infected socket
* Ant socket with wall defect.
* Pregnency
* Local or systemic conditions that will interfere with bone healing (uncontrolled diabetes mellitus or human immune deficiency virus infections, resonance therapy), bone disorders (hyperparathyroidism, osteoporosis, or Paget's disease.
* Patients who had subjected to intravenous and/or oral bisphosphonate therapy.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in implant stability | Baseline and after 6 month
  Implant stability will be assessed by using ( AnyCheck - Implant Stability Tester ) Utilizes physical tapping technique and dumping capacity analysis to measure implant stability with precision

SECONDARY OUTCOMES:
Change in marginal bone level and bone density around implants | Baseline and after 6 month
  To evaluate the amount of marginal bone loss and bone density around osseointegrated implants, all patient will be subjected to Cone beam computed tomography (CBCT) immediate postoperative and after 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Alaa Lecturer of OMFS, Study Director — faculty of Dental medicine Al-Azhar University
Locations (1):
- Faculty of dental medicine Al-Azhar university, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided